CLINICAL TRIAL: NCT05045391
Title: Prevalence of Chronic Pulmonary Aspergillosis and Antifungal Drug Resistance of Aspergillus Spp. in Pulmonary Tuberculosis Patients in Uzbekistan
Brief Title: Pulmonary Aspergillosis in Tuberculosis Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Research Institute of Epidemiology, Microbiology and Infectious Diseases, Uzbekistan (Other Government)
Responsible Party: Principal Investigator, Svetlana Osipova, MD, PhD, DS, Head of laboratory of immunology of parasitic and fungal diseases, Research Institute of Epidemiology, Microbiology and Infectious Diseases, Uzbekistan
Other Study IDs: 1/2021
Record Dates: First submitted 2021-09-06; First posted 2021-09-16 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Tuberculoses; Aspergillosis; Old Tuberculosis; Active Tuberculosis; Chronic Pulmonary Aspergillosis
MeSH Terms: conditions — Tuberculosis, Pulmonary; Aspergillosis; Latent Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- pulmonary tuberculosis (smear-positive) patients: Patients with pulmonary tuberculosis (smear-positive). Diagnosis of chronic pulmonary aspergillosis among patients with pulmonary tuberculosis (smear-positive)
  Interventions: Diagnostic Test: Aspergillus IgG detection
- pulmonary tuberculosis (smear-negative) patients: Patients with pulmonary tuberculosis (smear-positive). Diagnosis of chronic pulmonary aspergillosis among patients with pulmonary tuberculosis (smear-negative)
  Interventions: Diagnostic Test: Aspergillus IgG detection

INTERVENTIONS:
Diagnostic Test: Aspergillus IgG detection — Aspergillus IgG will be detected among pulmonary tuberculosis patients. 5 ml of vein blood will be collected for ELISA.
  Other Names: Mycological analysis of sputum

SUMMARY:
Pulmonary tuberculosis (PTB) is the most common cause of lung destruction, contributing to coinfections development, and Aspergillosis spp. is one of the most important. Diagnosis of chronic pulmonary aspergillosis (CPA) in PTB patients is difficult due to similarity of clinical and radiological data, especially in resource-constrained settings. Differentiation of PTB patients with singling out a group with a higher Aspergillus IgG level during the initial examination will help physicians to orient to further examination of CPA.

Objectives: to determine the prevalence of aspergillosis in Koch's bacillus-positive and Koch's bacillus-negative PTB patients and antifungal resistance of Aspergillus species isolates in Central Asia countries.

DETAILED DESCRIPTION:
Chronic pulmonary aspergillosis (CPA) complicates treated pulmonary tuberculosis (PTB), with high 5-year mortality. PTB affected an estimated 10.4 million people in 2016. Just 57% of PTB cases reported to the World Health Organization (WHO) were bacteriologically confirmed. CPA both complicates and mimics treated PTB. The prevalence of CPA in patients with treated TB and the contribution of misdiagnosed CPA to PTB prevalence estimates are unclear.

Mycological analysis of sputum for Aspergillus is often negative in CPA. Detection of Aspergillus IgG is one of the main analysis in CPA diagnosis, but until recently had been inadequately validated for use in this context. Both tests are infrequently available in areas of high PTB prevalence.

Antifungal therapy improves survival. But, survival rates vary significantly among published studies. Reported survival rates are 58%-93% at 1 year of follow-up, 17.5%-85% at 5 years of follow-up, and 30%-50% at 10 years of follow-up. In a selected group of patients with CPA, weekly subcutaneous injections of IFNγ has been shown to improve disease control and also helps with bacterial clearance. Several factors have been reported to affect mortality, including by underlying pulmonary disease, advanced age, NTM infection, quality of life scores, and serum albumin levels. No data on the prevalence of CPA among patients with PTB and resistance of Aspergillus spp. to antifungal drugs in Uzbekistan and neighboring countries.

The aim of the study is to determine the prevalence of aspergillosis in Koch's bacillus-positive and Koch's bacillus-negative PTB patients and antifungal resistance of Aspergillus species isolates in Central Asia countries.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary tuberculosis patients (smear-positive)
* Pulmonary tuberculosis patients (smear - negative)

Exclusion Criteria:

* neutropenia
* severe immunosuppression caused by cancer chemotherapy
* hematopoietic stem cell or solid organ transplantation
* HIV infected individuals

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pulmonary tuberculosis patients (smear-positive and smear - negative).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Aspergillus IgG | 2020-2025
  ELISA of serum of pulmonary tuberculosis patients.
Aspergillus sp. | 2020-2025
  Isolation of Aspergillus sp. among pulmonary tuberculosis patients
Antimicrobial resistance | 2020-2025
  Detection of antimicrobial resistance of fungi

CONTACTS AND LOCATIONS:
Overall Officials: Abdurakhim Toychiev, MD, PhD, Principal Investigator — Research institute of epidemiology, microbiology and infectious diseases
Locations (1):
- Research institute of epidemiology, microbiology and infectious diseases, Tashkent, Uchtepa, Uzbekistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Toychiev A, Belotserkovets V, Ignat'ev N, Madrakhimov S, Shaislamova M, Osipova S. Prevalence of chronic pulmonary aspergillosis and the antifungal drug resistance of Aspergillusspp. in pulmonary tuberculosis patients in Uzbekistan. Trop Doct. 2022 Oct;52(4):515-521. doi: 10.1177/00494755221110678. Epub 2022 Jun 30. PMID 35770798